CLINICAL TRIAL: NCT07019493
Title: Young Stroke Service Deep Phenotyping: Exploring Recovery in Young Adult Survivors of Stroke
Status: Not yet recruiting | Type: Observational
Sponsor: The Florey Institute of Neuroscience and Mental Health (Other)
Collaborators: University of Melbourne (Other); University of Newcastle, Australia (Other); Austin Health (Other Government); La Trobe University (Other); The Alfred (Other)
Responsible Party: Sponsor
Other Study IDs: Protocol One YSSDP; RARUR000042 (Other Grant/Funding Number: Medical Research Future Fund (Australia))
Record Dates: First submitted 2025-05-30; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Stroke Patients; Stroke; Stroke; Sequelae; Young Adults
Keywords: recovery; young stroke; ischemic stroke; hemorrhagic stroke; poststroke fatigue; post-stroke cognitive impairment; function; mood
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young adult stroke survivors (age 18 to 55 inclusive)
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — Not applicable: Observational cohort study

SUMMARY:
We are running a small, early-phase research study across several hospitals in Melbourne, Australia. The study will involve up to 100 young adults between the ages of 18 and 55 who have had a stroke. Our goal is to test how practical it is to carry out a detailed health assessment process-called "deep phenotyping"-with this group.

This process involves collecting a wide range of information and samples from stroke survivors to better understand each participant's condition. We'll look at how well this approach works in practice, including how easy it is to use, whether it's done consistently, and how acceptable it is to participants.

At the same time, we'll also explore how different factors-such as biological markers (biomarkers), age, sex, type of stroke, lifestyle, and environment-might be related to stroke recovery. This pilot study will help us prepare for larger studies in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 55 years.
2. Within one month of acute stroke confirmed with standard of care brain imaging or clinical diagnosis

Exclusion Criteria:

1. Severe, intercurrent or progressive illness likely to EITHER

   1. Have a prognosis for survival under 24 months; OR
   2. In the opinion of the investigator will mask the importance to the individual participant data (e.g. severe MS, dementia, etc)
2. Major psychiatric condition requiring medical intervention

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young adult stroke survivors within 1 month of stroke
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Implementability (feasibility, fidelity and acceptability) | From enrolment to the six month assessment visit
  Evaluation of the implementability will include assessment of the protocol's:
  * Feasibility, e.g.
    * Recruitment rate
    * Retention
    * Proportion of participants screened that enrolled
    * Safety via adverse events
  * Fidelity, e.g.
    * Proportion of assessments attended
    * Proportion of data collected and biobanked or analysed
  * Acceptability, e.g. o Participant acceptability surveys

SECONDARY OUTCOMES:
Fatigue Severity Scale | 6 months
  FSS: A 9-item (or 7-item with the first two items removed) measure of fatigue impairment.
  Measured at baseline (<1month post stroke), 3- and 6-months post stroke.
Visual Analogue Scale to Assess Fatigue (VAS-F) | Assessment at <1, 3- and 6-months post stroke
  18-item visual analogue scale of fatigue and energy items.
Modified Fatigue Impact Scale (MFIS) is a multidimensional scale that reports physical, psychological and cognitive aspects of fatigue | 6 months
  A multidimensional 21-item measure that evaluates physical, psychological and cognitive aspects of fatigue. Measured at baseline (<1month post stroke), 3- and 6-months post stroke.
Cognitive Assessment | 6 months
  Assessment to evaluate cognitive domains such as visuospatial memory, auditory verbal learning, visual attention, task switching, verbal fluency, and verbal short-term and working memory. Assessment <1-month, 3- and 6-months post stroke.
modified Rankin Scale (mRS) | 6 months
  Single-item evaluation of global disability. Assessed at <1-month, 3- and 6-months post stroke
10 metre walk test (10mWT) | 6 months
  Gait assessment, evaluated <1-month, 3- and 6-months post stroke
Visual Analogue Scale of the Impact of Fatigue on Communication Ability | 6 months
  Visual analogue scale (0-10) assessing the impact of fatigue on communication ability.
  Measured at baseline (<1month post stroke), 3- and 6-months post stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Thijs, MD, PhD, Principal Investigator — Florey Institute of Neuroscience and Mental Health
Locations (1):
- Florey Institute of Neuroscience and Mental Health, Melbourne Brain Centre, Heidelberg, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided
Sharing of individual patient data will be considered upon reasonable request by qualified researchers with appropriate IRB/HREC approval